CLINICAL TRIAL: NCT00482287
Title: A Phase II, Randomized, Double Blind, Placebo-controlled, Dose-escalating Study to Assess the Pharmacokinetics and Pharmacodynamics of MTR105 in Cardiac Surgery Induced Hypotension Patients During Weaning Off Cardiopulmonary Bypass
Brief Title: Pharmacokinetics and Pharmacodynamics of MTR105 in Hypotensive Cardiac Surgery Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Site did not recruit any patients
Sponsor: Meditor Pharmaceuticals Ltd. (Industry)
Responsible Party: Adrian Harel, Meditor Pharmaceuticals Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTR-105-US-102
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hypotension; Cardiopulmonary Bypass
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Other): Dose level 0.3 mg/kg with 6 active and 2 placebo
  Interventions: Drug: MTR105
- 2 (Other): Dose level 0.6 mg/kg 6 patients active and 2 placebo
  Interventions: Drug: MTR105
- 3 (Other): Dose level 1.2 mg/kg 6 active and 2 placebo
  Interventions: Drug: MTR105
- 4 (Other): Dose level 2.4 mg/kg 6 active and 2 placebo
  Interventions: Drug: MTR105

INTERVENTIONS:
Drug: MTR105 — Intravenous administration, dose escalating (4 arms), single dose

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetic and the pharmacodynamic effects of escalating doses of MTR105 while weaning from bypass in a hypotensive population of cardiac surgery patients.

DETAILED DESCRIPTION:
The study is a prospective, randomized, four-arm, dose-escalating, double blind, placebo controlled study evaluating the safety, pharmacokinetics, and pharmacodynamics of four dose levels of MTR105 in patients undergoing cardiac surgery utilizing cardiopulmonary bypass presenting hypotension upon weaning off bypass.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 years or older
* Referred for cardiac surgery requiring the use of CPB.
* Elective or urgent surgeries (non emergency operations).
* LVEF ≥40 based on cardiac catheterization results
* Normal renal function at study entry
* Normal hepatic function (within normal laboratory ranges) at study entry
* Normal coagulation status at study entry as judged by PT, PTT, fibrinogen and platelet count.
* Willingness to participate in the study and adhere to the study design.
* Willingness to sign an informed consent form.

Exclusion Criteria:

* Emergency operation
* Pulmonary hypertension (PA systolic pressure >60 mmHg)
* Ejection fraction less than 35% during weaning from bypass or cardiac index of less than 1.8
* Neurological events such as prior CVA, TIA or symptomatic carotid stenosis within 1 year of presenting for surgery
* Body weight <40 Kg
* Pregnancy
* Malignancy within 1 year of presenting for surgery
* Systemic infection as evidenced by elevated WBC or fever >38.5 C
* Usage of vasoactive medications within 24 hours except short term use of a vasoconstrictor during induction.
* Participation in any other investigational drug or device study within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Hemodynamic parameters | 24 hours

SECONDARY OUTCOMES:
Pharmacokinetics | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Penny Sappington, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States